CLINICAL TRIAL: NCT02748135
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation Study of TB-403 in Pediatric Subjects With Relapsed or Refractory Medulloblastoma, Neuroblastoma, Ewing Sarcoma or Alveolar Rhabdomyosarcoma
Brief Title: A Study of TB-403 in Pediatric Subjects With Relapsed or Refractory Medulloblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncurious NV (Industry)
Collaborators: Beat Childhood Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-403-001
Record Dates: First submitted 2016-04-08; First posted 2016-04-22 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Relapsed or Refractory Medulloblastoma (MB), Neuroblastoma (NB), Ewing Sarcoma (ES) and Alveolar Rhabdomyosarcoma (ARMS)
MeSH Terms: conditions — Recurrence; Medulloblastoma; Neuroblastoma; Sarcoma, Ewing; Rhabdomyosarcoma, Alveolar | interventions — TB-403

ARMS (4):
- TB-403 20mg/kg (Experimental)
  Interventions: Drug: TB-403 20mg/kg
- TB-403 50mg/kg (Experimental)
  Interventions: Drug: TB-403 50mg/kg
- TB-403 100mg/kg (Experimental)
  Interventions: Drug: TB-403 100mg/kg
- TB-403 175mg/kg (Experimental)
  Interventions: Drug: TB-403 175mg/kg

INTERVENTIONS:
Drug: TB-403 20mg/kg — bi-weekly intravenous doses of TB-403 20mg/kg
  Arms: TB-403 20mg/kg
Drug: TB-403 50mg/kg — bi-weekly intravenous doses of TB-403 50mg/kg
  Arms: TB-403 50mg/kg
Drug: TB-403 100mg/kg — bi-weekly intravenous doses of TB-403 100mg/kg
  Arms: TB-403 100mg/kg
Drug: TB-403 175mg/kg — bi-weekly intravenous doses of TB-403 175mg/kg
  Arms: TB-403 175mg/kg

SUMMARY:
The purpose of this study is to assess the safety and tolerability profile of TB-403 (humanized monoclonal antibody against placental growth factor (PlGF)) in pediatric subjects with relapsed or refractory Medulloblastoma.

DETAILED DESCRIPTION:
The maximum tolerated dose of TB-403 will be determined in pediatric subjects with relapsed or refractory Medulloblastoma (MB) and as well Neuroblastoma (NB), Ewing Sarcoma (ES) and Alveolar Rhabdomyosarcoma (ARMS).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent (Subject or legal representative)
2. Be > 6 months and < 18 years of age. For each dose cohort, the first 3 subjects must be at least 2 years of age
3. Have a histologically-confirmed diagnosis of MB, NB, ES, or ARMS
4. Have documented relapse or refractoriness after standard-of-care therapy
5. Have undergone magnetic resonance imaging (MRI) for MB (brain [all cohorts] and spinal cord [cohort 4 only], a computerized tomography (CT) / metaiodobenzylguanidine (MIBG) scan for NB, and CT / magnetic resonance imaging (MRI) for ES or ARMS within 1 month prior to first dose of study treatment
6. Have a Lansky score ≥ 40 for subjects up to 16 years of age or a Karnofsky score ≥ 40 for subjects 16 years of age to < 18 years
7. Have adequate organ function, defined as:

   * Peripheral absolute neutrophil count ≥ 1.5 × 10^9/L
   * Platelet count ≥ 100 × 10^9/L (transfusion to reach this level is permitted)
   * Hemoglobin ≥ 8mg/dL (transfusion to reach this level is permitted)
   * International normalized ratio (INR) < 1.5; partial thromboplastin time (PTT) < 1.5 upper limit of normal (ULN)
   * Creatinine clearance > 50mL/min/1.73m2 or serum creatinine ≤ specified maximum values based on age, as described below:
   * 6 months to 3 years of age: serum creatinine ≤ 0.4mg/dL
   * 3 to 13 years of age: serum creatinine ≤ 0.7mg/dL
   * > 13 years of age: serum creatinine ≤ 1mg/dL
   * Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) < 2.5 × ULN; serum bilirubin < 1.5 × ULN
8. Have no symptoms of cranial hypertension or convulsions within 14 days before Cycle 1 Day 1 (anti-epileptic drugs and corticoids are allowed to control any preexisting symptoms)
9. If female of child bearing potential, must not be lactating and must have a negative pregnancy test (blood or urine, at the discretion of the investigator) prior to enrollment and use effective contraception during study participation. Women should continue effective contraception for 3 months following last dose of TB-403.
10. If a sexually-active male, must agree to use a latex condom during any sexual contact with females of child bearing potential while participating in the study and for 3 months following last dose of TB-403.
11. For subjects on corticosteroids for endocrine deficiencies or tumor-associated symptoms, must be on a stable (or decreasing) dose for at least 7 days before first dose of study treatment.

Exclusion Criteria:

1. Have any clinically significant disease considered by the investigator to interfere with study participation
2. Have not fully recovered from the acute toxic effects of prior anticancer therapy (e.g., chemotherapy, immunotherapy, radiation therapy) or are currently receiving cytotoxic chemotherapy, immunotherapy or radiation therapy. Subjects must be within the following timelines relative to first dose of study treatment:

   * Myelosuppressive chemotherapy: Must not have received within 2 weeks (6 weeks if prior nitrosourea)
   * Hematopoietic growth factors: At least 5 days since the completion of therapy with a growth factor
   * Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the Sponsor
   * Immunotherapy: At least 6 weeks since the completion of any type of immunotherapy, e.g., tumor vaccines
   * Monoclonal antibodies: At least 7 days or 3 half-lives, whichever is longer, must have elapsed since prior treatment with a monoclonal antibody
   * Radiotherapy: At least 14 days since the last treatment except for radiation delivered with palliative intent to a non-target site
   * Stem Cell Transplant or Rescue: No evidence of active graft vs. host disease and ≥ 2 months must have elapsed since transplant
3. Have participated in another therapeutic clinical trial with an investigational drug within 1 month before first dose of study treatment
4. Have any known active uncontrolled infection
5. Have had major surgery or bone fracture within 28 days before first dose of study treatment
6. Have previously received TB-403
7. Have a history of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational drug
8. Are receiving increasing doses of corticosteroids
9. Are eligible for a curative treatment option
10. Have had a prior thrombotic event (e.g., pulmonary embolism, deep vein thrombosis) or are currently receiving therapeutic or prophylactic doses of anticoagulants.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05; Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint will be the determination of the maximum tolerated dose (MTD) / study maximum dose (SMD) based on the occurrence of dose-limiting toxicities (DLTs) during the 28-day DLT assessment period. | Day28

SECONDARY OUTCOMES:
TB-403 total exposure (AUC∞) after single ascending dose | Day 1, day 4, day 8, day 15, day 29, day 60, day 90, day 165 and day 195.
TB-403 Dose/CL after single ascending dose | Day 1, day 4, day 8, day 15, day 29, day 60, day 90, day 165 and day 195.
TB-403 Volume of the central compartment (Vc) after single ascending dose | Day 1, day 4, day 8, day 15, day 29, day 60, day 90, day 165 and day 195.
TB-403 Volume of distribution at steady-state (Vss) after single ascending dose | Day 1, day 4, day 8, day 15, day 29, day 60, day 90, day 165 and day 195.
TB-403 terminal half-life (t½,z) after single ascending dose | Day 1, day 4, day 8, day 15, day 29, day 60, day 90, day 165 and day 195.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Little Rock, Arkansas
  - Oakland, California
  - Hartford, Connecticut
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - St Louis, Missouri
  - Hackensack, New Jersey
  - Charleston, South Carolina
  - Austin, Texas
  - Dallas, Texas